CLINICAL TRIAL: NCT05499806
Title: Cohort Study on the Effects of Aging in Acquired Brain Injury Patients
Acronym: BRAINReADAPT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Medical Center Groningen (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Joukje van der Naalt, Prof. dr. J. van der Naalt, University Medical Center Groningen
Other Study IDs: NL79072.042.21
Record Dates: First submitted 2022-07-26; First posted 2022-08-12 (Actual); Last update posted 2022-08-12 (Actual); Status verified 2022-08

CONDITIONS: Acquired Brain Injury; Subarachnoid Hemorrhage; Traumatic Brain Injury; Cerebrovascular Accident
MeSH Terms: conditions — Brain Injuries; Subarachnoid Hemorrhage; Brain Injuries, Traumatic; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Acquired Brain Injury Patients: Questionnaire and, if the requirements are met, a neuropsychological assessment.
- Healthy volunteers: Questionnaire and, if the requirements are met, a neuropsychological assessment.

SUMMARY:
A prospective cohort study (questionnaires), with an embedded case control study (neuropsychological assessments) in which the data is gathered within a timeframe of 3 years. A group of 700 patients and a group of 100 healthy volunteers will be participating.

DETAILED DESCRIPTION:
In the Netherlands an estimated 650.000 people live with the daily consequences of an Acquired Brain Injury (ABI). A substantial amount of these patients acquired their brain injury (traumatic brain injury, subarachnoid hemorrhage or cerebrovascular accident) at a relatively young age: between 18 and 50 years old. The chain-of-care for ABI aims for recovery in the subacute phase, usually within a period of one year after injury. After an adaptation period, the patients reach a new balance, with stabilization of complaints and reintegration, sometimes with the necessity of modifications. The group of patients who acquired a brain injury at a young age, have to face the effects of aging like decreased cognitive functions, which can cause the participation level to drop. This is called the ABI-effect in the current study. At this moment, insufficient information is available about the functioning of people who suffered ABI multiple years ago and have established a new balance, and now make the transition to an older phase of live.

Primary objective:

Explore the prevalence of the ABI-effect, by mapping the participation level.

Secondary objective:

Substantiate the occurence of the ABI-effect, by mapping cognitive functions of patients and compare these to healthy controls.

Tertiary objective:

Gain insight in the need of care for patients, to enhance regular care after ABI.

ELIGIBILITY:
Inclusion Criteria:

* Current age range between 50-67 years [Rationale: having an age that enables the patient to experience the effects of aging with a low risk of neurodegenerative disease]
* Able to complete questionnaires independently

Additionally, patients must also meet the following criteria:

* Age of acquiring the ABI ≧ 25 years [Rationale: the brain is supposed to be fully developed at a maximum capacity
* ABI must be ≧ 5 years ago] [Rationale :time period regarded sufficient to have achieved a stable level of cognitive functioning and participation after an ABI]
* ABI diagnosis at hospital admission with abnormalities at the brain-CT or MRI
* Independent regarding Activities of Daily Living
* Not living in a long-term care facility

Exclusion Criteria:

* Psychiatric disease (for which participant is currently treated)
* Accompanying disease with reduced life expectancy
* Neurological disease (including recurrent ABI for patients)
* Language barriers prohibiting and completion of Dutch questionnaires
* Alcohol or drug abuse
* Suspected neurodegenerative disease

Ages: 50 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who have suffered an acute ABI defined by a traumatic brain injury, stroke or subarachnoid haemorrhage who have been admitted at the UMCG or one of the other participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2022-03-18 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of the ABI-effect | A minimum of 5 years after ABI
  The percentage of patients experiencing the ABI-effect. Also, a 95% confidence interval of this prevalence will be calculated.

SECONDARY OUTCOMES:
Cognitive functions of patients and healthy volunteers | A minimum of 5 years after ABI for patients
  The significant difference in cognitive functions between the patient groep and the healthy controls

CONTACTS AND LOCATIONS:
Locations (2):
- Netherlands (2):
  - Isala klinieken, Zwolle, Overijssel
  - Revalidatiecentrum Heliomare Wijk aan Zee, Wijk aan Zee

IPD SHARING:
Plan to Share IPD: No